CLINICAL TRIAL: NCT03205917
Title: A Phase 1 Randomized Placebo-controlled Clinical Trial of the Safety, Pharmacokinetics and Antiviral Activity of PGDM1400 and PGT121 and VRC07-523LS Monoclonal Antibodies in HIV-uninfected and HIV-infected Adults
Brief Title: A Clinical Trial of PGDM1400 and PGT121 and VRC07-523LS Monoclonal Antibodies in HIV-infected and HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Beth Israel Deaconess Medical Center (Other); Ragon Institute of MGH, MIT and Harvard (Other); University of Texas Health, Houston AIDS Research Team (HART) (Unknown); Orlando Immunology Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAVI T002
Record Dates: First submitted 2017-05-12; First posted 2017-07-02 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1A HIV-Uninfected (Experimental): PGDM1400 low dose
  Interventions: Biological: PGDM1400/Placebo (3mg/kg IV)
- Group 1B HIV-Uninfected (Experimental): PGDM1400 mid dose
  Interventions: Biological: PGDM1400/Placebo (10mg/kg IV)
- Group 1C HIV-Uninfected (Experimental): PGDM1400 high dose
  Interventions: Biological: PGDM1400/Placebo (30mg/kg IV)
- Group 2A HIV-Uninfected (Experimental): PGDM1400 + PGT121 low dose
  Interventions: Biological: PGDM1400 + PGT121/Placebo (3mg/kg + 3mg/kg IV)
- Group 2B HIV-Uninfected (Experimental): PGDM1400 + PGT121 mid dose
  Interventions: Biological: PGDM1400 + PGT121/Placebo (10mg/kg + 10mg/kg IV)
- Group 2C HIV-Uninfected (Experimental): PGDM1400 + PGT121 high dose
  Interventions: Biological: PGDM1400 + PGT121/Placebo (30mg/kg + 30mg/kg IV)
- Group 3A HIV-infected off ART (Experimental): PGDM1400 + PGT121 + VRC07-523LS at 20mg/kg; HIV+ without ART
  Interventions: Biological: PGDM1400 + PGT121 + VRC07-523LS (20mg/kg + 20mg/kg + 20 mg/kg IV)
- Group 3B HIV-infected off ART (Experimental): PGDM1400 + PGT121 at high dose; HIV + without ART
  Interventions: Biological: PGDM1400 + PGT121 (MTD IV)

INTERVENTIONS:
Biological: PGDM1400/Placebo (3mg/kg IV) — 3/1 (6/2 if DLT)
  Arms: Group 1A HIV-Uninfected
Biological: PGDM1400/Placebo (10mg/kg IV) — 3/1 (6/2 if DLT)
  Arms: Group 1B HIV-Uninfected
Biological: PGDM1400/Placebo (30mg/kg IV) — 3/1 (6/2 if DLT)
  Arms: Group 1C HIV-Uninfected
Biological: PGDM1400 + PGT121/Placebo (3mg/kg + 3mg/kg IV) — 3/1 (6/2 if DLT)
  Arms: Group 2A HIV-Uninfected
Biological: PGDM1400 + PGT121/Placebo (10mg/kg + 10mg/kg IV) — 3/1 (6/2 if DLT);
  Arms: Group 2B HIV-Uninfected
Biological: PGDM1400 + PGT121/Placebo (30mg/kg + 30mg/kg IV) — 3/1 (6/2 if DLT)
  Arms: Group 2C HIV-Uninfected
Biological: PGDM1400 + PGT121 + VRC07-523LS (20mg/kg + 20mg/kg + 20 mg/kg IV) — 3 (max 9)
  Arms: Group 3A HIV-infected off ART
Biological: PGDM1400 + PGT121 (MTD IV) — 3 (max 9)
  Arms: Group 3B HIV-infected off ART

SUMMARY:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics and anti-viral efficacy of the PGDM1400 and PGT121 and VRC07-523LS mAbs for HIV prevention and therapy.

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safety, tolerability, pharmacokinetics and anti-viral efficacy of the PGDM1400, PGT121 and VRC07-523LS mAbs for HIV prevention and therapy. PGDM1400, PGT121 and VRC07-523LS mAbs are recombinant human IgG1 monoclonal antibodies that target V1V2 (PGDM1400), a V3 glycan-dependent epitope (PGT121) and the CD4 binding site (VRC07-523LS) epitope region of the HIV envelope protein. PGT121, PGDM1400 and VRC07-523LS mAb were chosen for this study because of their potency, their ability to neutralize a wide array of cross-clade HIV viruses in a complementary pattern and their proven antiviral activity in animal studies e.g., their capacity to robustly prevent and treat simian-human immunodeficiency virus (SHIV) in rhesus monkeys.

ELIGIBILITY:
Groups 1 and 2 Inclusion Criteria:

* HIV-uninfected males or females age 18-50 years old
* Willing to maintain low risk behavior for HIV infection

Groups 1 and 2 Exclusion Criteria:

• Confirmed HIV-infection, pregnancy or lactation, significant acute or chronic disease and clinically significant laboratory abnormalities

Group 3 Inclusion Criteria:

* HIV-infected males or females age 18-65 years old
* Not on antiretroviral therapy with HIV-1 RNA plasma level between 1,000 and 100,000 copies/ml, CD4 cell count ≥ 300 cells/uL

Group 3 Exclusion Criteria:

• Significant acute or chronic medical condition other than HIV infection, and clinically significant laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 Months post infusion
  1. Proportion of participants with moderate or greater reactogenicity (e.g., solicited adverse events) for 3 days following IV infusion of PGDM1400 mAb alone, and a combination of PGDM1400 mAb and PGT121 mAb, and a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb
  2. Proportion of participants with adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, during the first 56 days following IV infusion of PGDM1400 mAb alone and a combination of PGDM1400 mAb and PGT121 mAb, and a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb, that are moderate or greater, and/or related to PGDM1400 mAb or PGT121 mAb or VRC07-523LS mAb
  3. Proportion of participants with SAEs throughout the study period following IV infusion of PGDM1400 mAb alone and a combination of PGDM1400 mAb and PGT121 mAb, and a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb, that are related to PGDM1400 mAb or PGT121 mAb or VRC07-523LS mAb
Elimination half-life (t1/2) | 6 Months post infusion
  Elimination half-life following IV infusion of PGDM1400 mAb alone or a combination of PGDM1400 mAb and PGT121 mAb in HIV-uninfected and HIV-infected adults; or a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb in HIV-infected adults
Clearance (CL/F) | 6 months post infusion
  Clearance following IV infusion of PGDM1400 mAb alone or a combination of PGDM1400 mAb and PGT121 mAb in HIV-uninfected and HIV-infected adults; or a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb in HIV-infected adults.
Volume of distribution (Vz/F) | 6 months post infusion
  Volume of distribution following IV infusion of PGDM1400 mAb alone or a combination of PGDM1400 mAb and PGT121 mAb in HIV-uninfected and HIV-infected adults; or a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb in HIV-infected adults
Area under the concentration decay curve (AUC) | 6 months post infusion
  AUC following IV infusion of PGDM1400 mAb alone or a combination of PGDM1400 mAb and PGT121 mAb in HIV-uninfected and HIV-infected adults; or a combination of PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb in HIV-infected adults
Impact of viral load and/or ART | 6 months post infusion
  Impact of viral load and/or ART on PGDM1400 mAb and PGT121 mAb and VRC07-523LS mAb disposition
Antiviral activity of PGDM1400 in combination with PGT121 or PGDM1400 in combination with PGT121 and VRC07-523LS mAbs | 6 Months post infusion
  Antiviral activity following IV infusion of PGDM1400 mAb in combination with PGT121 mAb, or PGDM1400 mAb in combination with PGT121 mAb and VRC07-523LS mAb, in viremic HIV-infected adults not on ART:
  Change in plasma HIV-1 RNA levels from baseline (mean of pre-entry and entry values)

SECONDARY OUTCOMES:
Serum antibody titers against bNAbs | 6 Months post infusion
  Serum anti-PGDM1400 antibody titers, Serum anti-PGT121 antibody titers and Serum anti-VRC07-523LS antibody titers
CD4+ T cell count | 6 Months post infusion
  Determine if IV infusion of PGDM1400 mAb in combination with PGT121 mAb, or PGDM1400 mAb in combination with PGT121 mAb and VRC07-523LS mAb, has any impact on CD4+ T cell counts in HIV-infected adults. Change in CD4+ T cell count compared to baseline as measured by single platform flow cytometry
HIV genotyping of circulating virus | 6 Months post infusion
  Compare plasma virus genotype activity before and after IV infusion of PGDM1400 mAb in combination with PGT121 mAb, or PGDM1400 mAb in combination with PGT121 mAb and VRC07-523LS mAb to determine if PGDM1400 mAb and PGT121 mAb and/or PGT121VRC07-523LS mAb induced viral escape mutations have developed in viremic HIV-infected adults not on ART
  Genotypic analysis: Development of sequence variations in epitopes known to result in reduced PGDM1400 mAb and/or PGT121 mAb and/or VRC07-523LS mAb neutralization susceptibility or known to cause resistance to antiretroviral drugs
HIV phenotyping of circulating virus | 6 months post infusion
  Compare plasma virus phenotypic activity before and after IV infusion of PGDM1400 mAb in combination with PGT121 mAb, or PGDM1400 mAb in combination with PGT121 mAb and VRC07-523LS mAb to determine if PGDM1400 mAb and PGT121 mAb and/or PGT121VRC07-523LS mAb induced viral escape mutations have developed in viremic HIV-infected adults not on ART. Phenotypic analysis: Changes in viral susceptibility to PGDM1400 mAb and/or PGT121 mAb and/or VRC07-523LS mAb neutralization
  Phenotypic analysis: Changes in viral susceptibility to PGDM1400 mAb and/or PGT121 mAb and/or VRC07-523LS mAb neutralization.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Juelg, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center, Center for Virology and Vaccine Research, Ragon Institute of MGH, MIT and Harvard; Kathryn Stephenson, MD, MPH, Study Chair — Beth Israel Deaconess Medical Center, Center for Virology and Vaccine Research
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Julg B, Stephenson KE, Wagh K, Tan SC, Zash R, Walsh S, Ansel J, Kanjilal D, Nkolola J, Walker-Sperling VEK, Ophel J, Yanosick K, Borducchi EN, Maxfield L, Abbink P, Peter L, Yates NL, Wesley MS, Hassell T, Gelderblom HC, deCamp A, Mayer BT, Sato A, Gerber MW, Giorgi EE, Gama L, Koup RA, Mascola JR, Monczor A, Lupo S, Rolle CP, Arduino R, DeJesus E, Tomaras GD, Seaman MS, Korber B, Barouch DH. Safety and antiviral activity of triple combination broadly neutralizing monoclonal antibody therapy against HIV-1: a phase 1 clinical trial. Nat Med. 2022 Jun;28(6):1288-1296. doi: 10.1038/s41591-022-01815-1. Epub 2022 May 12. PMID 35551291
- See also: IAVI Website — http://iavi.org